CLINICAL TRIAL: NCT02271152
Title: Focal Electrical Source and Trigger Mapping During Atrial Fibrillation
Brief Title: FAST Mapping During Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Vijay Chauhan, Cardiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-121
Record Dates: First submitted 2014-10-18; First posted 2014-10-22 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAST ablation + PVI (Experimental): FAST mapping and ablation will be performed in addition to PVI
  Interventions: Procedure: FAST mapping and ablation; Procedure: PVI
- PVI (Active Comparator): Pulnonary vein isolation will be performed
  Interventions: Procedure: PVI

INTERVENTIONS:
Procedure: FAST mapping and ablation
  Arms: FAST ablation + PVI
Procedure: PVI

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia worldwide with a prevalence of 8% in the elderly. AF is responsible for frequent hospitalizations, stroke, heart failure and mortality. AF catheter ablation is an important treatment strategy for patients suffering from AF, but the success rate remains low after conventional pulmonary vein isolation (PVI). The mechanism perpetuating AF is poorly understood. Focal electrical sources and triggers (FAST) may sustain AF in some patients, which makes them a potential therapeutic target for ablation. However, finding FAST is very challenging due to complex nature of AF electrical signals. In this study, the investigators will attempt to localize focal electrical sources and triggers (FAST mapping) in patients undergoing AF ablation using custom software that evaluates periodicity and waveform morphology. Patients will be randomized to one of two AF ablation strategies, namely FAST mapping/ablation + PVI vs. PVI alone. The investigators will determine which strategy leads to better clinical outcome postablation.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be over the age 18 and have a clinical indication for their first catheter ablation of AF because of symptomatic AF.
* This will include patients with either high burden paroxysmal (>4 self-terminating episodes of AF within the last 6 months with two episodes lasting at least 6 hours within the last year) or persistent AF (lasting ≥7 days, but which can still be converted to sinus rhythm).

Exclusion Criteria:

* The major exclusion criteria will include:

  * long-standing persistent AF (ie. AF which cannot be converted to sinus rhythm, or where multiple attempts at restoring sinus rhythm have failed)
  * rheumatic valvular disease
  * hypertrophic cardiomyopathy
  * uncorrected cardiac shunts (eg. secundum ASD)
  * severe mitral regurgitation or mechanical mitral valve
  * left atrial size >55 mm (echo derived parasternal long axis view).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Time to first symptomatic atrial fibrillation recurrence postablation | 3 months postablation

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada